CLINICAL TRIAL: NCT01344980
Title: A Pilot Study of a Randomized Controlled Trial Comparing Stainless Steel Suture Repair Coupled With Aggressive Post-Operative Rehabilitation to Polypropylene Suture Paired With Active Range of Motion Rehabilitation
Brief Title: The Effects of a Stainless Steel Suture MGH Flexor Tendon Repair Coupled With Early Aggressive Range of Motion Rehabilitation: a Randomized Controlled Trial
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Manitoba (Other)
Responsible Party: Ian MacArthur (principle investigator), University of Manitoba: Department of Surgery: Section of Plastic Surgery
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: B2010:119
Record Dates: First submitted 2011-04-28; First posted 2011-04-29 (Estimated); Last update posted 2011-04-29 (Estimated); Status verified 2011-02

CONDITIONS: Zone 2 Flexor Tendon Lacerations of the Hand

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Stainless steel MGH (Experimental): Patients in this study arm will have their flexor tendon laceration repaired using stainless steel suture (size 3-0) in an MGH repair technique. They will then undergo aggressive early active range of motion rehabilitation post-operatively.
  Interventions: Procedure: Stainless steel suture; Behavioral: Aggressive early active range of motion rehabilitation
- Polypropylene DOLL (Active Comparator): Patients in this study arm will have their flexor tendon laceration repaired using polypropylene suture (size 3-0) in a double-locking loop repair technique. They will then undergo aggressive early active range of motion rehabilitation post-operatively.
  Interventions: Procedure: Polypropylene suture; Behavioral: Early active range of motion rehabilitation

INTERVENTIONS:
Procedure: Stainless steel suture — Stainless steel suture material will be used (size 3-0) in an MGH repair technique
  Arms: Stainless steel MGH
Procedure: Polypropylene suture — Polypropylene suture (size 3-0) will be used in a double-locking loop repair technique
  Arms: Polypropylene DOLL
Behavioral: Aggressive early active range of motion rehabilitation — Patients undergoing this form of rehabilitation will have their splints discontinued at 4 weeks and ideally will be back at work at normal duties by 6 weeks. This rehabilitation uses more movement at a faster progression than other early active range of motion protocols.
  Arms: Stainless steel MGH
Behavioral: Early active range of motion rehabilitation — Patients undergoing this form of rehabilitation will have their splints discontinued at 6 weeks and ideally will be back at work at normal duties by 10-12 weeks. This rehabilitation uses less movement at a slower progression than the early AROM rehabilitation protocol specified in the experimental group
  Arms: Polypropylene DOLL

SUMMARY:
The investigators are comparing the combination of a stainless steel repair and aggressive early active range of motion rehabilitation protocol for flexor tendon lacerations in the hand with a current, accepted treatment offered at our institution. Outcomes to be assessed will be time to return to work, joint range of motion in the injured fingers, and any potential complications that may arise (ex: surgical infections or repair rupture). All proposed treatments included in this study are currently being offered at our institution, but not in a randomized fashion.

DETAILED DESCRIPTION:
This study will serve as a pilot-study for a future randomized controlled trial. Adult patients with zone 2 flexor tendon lacerations of the hand (anatomically from the A1 pulley of the hand to the insertion of the flexor digitorum superficialis) who have presented to the emergency room acutely (within 1 week of injury) at the Health Sciences Center in Winnipeg will be asked for their participation in this study. Consent will be obtained by a plastic surgery resident either in the emergency room or in the plastic surgency emergency decanting clinic. The investigators will include twenty-four patients in the study, randomized into one of two treatment groups (groups A and B) by block randomization. Randomization will be done once patients agree to participate in the study. All patients will be booked for surgery on the emergency slate. Each treatment group will be treated by a single surgeon who is an expert at treatment of these injuries. Group A patients will have their laceration(s) repaired using a modified Becker repair technique using stainless steel suture in the operating room, and then will proceed to undergo an aggressive early active range of motion rehabilitation administered by the hand therapists at HSC. Group B patients will undergo a double-locking loop suture repair using polypropylene. They will then undergo a less aggressive active range of motion rehabilitation protocol which is currently offered to patients at our center. Follow-up will occur in plastic surgery outpatient clinic at post-operative weeks 1, 2, 4, 6 and 12. Follow-up with hand therapy will be at the discretion of the therapists. At each visit with hand therapy, joint range of motion will be assessed at the PIP and DIP joints in the affected fingers. Final range of motion will be assessed using the Strickland system for evaluating flexor tendon surgery outcomes, and will be done by a blinded hand therapist.

ELIGIBILITY:
Inclusion Criteria:

* adults
* living in Winnipeg, Manitoba
* zone II flexor tendon lacerations in a single finger
* able to consent to and comply with surgery

Exclusion Criteria:

* crush injuries
* vascular injuries requiring re-vascularization
* fractures
* infection
* prior hand injury requiring surgery

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2011-06; Primary Completion 2012-06 (Estimated); Study Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
Return to work | Post-operative weeks 1, 2, 4, 6 and 12
  At each clinic visit at the above mentioned time periods, the clinician will ask the patient if they have returned to work (if applicable)
Finger joint range of motion (PIP, DIP, MCP) | Post-operative weeks 1, 2, 4, 6 and 12
  At each clinic / occupational therapy visit, a blinded assessor will determine the total range of motion of the finger DIP, PIP and MCP joints

SECONDARY OUTCOMES:
Compliance with therapy | Post-operative weeks 1, 2, 4, 6 and 12
  At each clinic and occupational therapy visit, an assessor will ask the patient if they have been compliant with therapy
Rupture | Post-operative weeks 1, 2, 4, 6 and 12
  At each follow-up visit with the clinician or occupational therapist, the presence of a rupture will be assessed for clinically. Alternatively this will be recorded if the patient presents to the emergency room with a flexor tendon rupture
Infection | Post-operative weeks 1, 2, 4, 6 and 12
  At each clinic visit, the patient will be assessed clinically for the presence or absence of an infection. This will also be noted if the patient presents to the emergency room.
Attendance with follow-up clinic and occupational therapy | Post-operative weeks 1, 2, 4, 6 and 12
  The patient's attendance will be determined at each clinic or occupational therapy visit.
Use of oral analgesics | Post-operative weeks 1, 2, 4, 6 and 12
  At each clinic visit, the patient will be asked if they are still using oral analgesics
Oral antibiotic usage | Post-operative weeks 1, 2, 4, 6 and 12
  At each clinic visit, the patient will be asked if they are using oral antibiotics.
Wound dehiscence (breakdown) | Post-operative weeks 1, 2, 4, 6 and 12
  At each clinic and occupational therapy visit, the patient will be assessed to determine if a wound dehiscence (breakdown) has occurred.
Use of occupational therapy adjunctive treatments | Post-operative weeks 1, 2, 4, 6 and 12
  At each occupational therapy visit, it will be recorded that they are either using or not using occupational therapy adjunctive treatments (ex: coban tape, ultrasound or electrical stimulation)

CONTACTS AND LOCATIONS:
Locations (1):
- Health Sciences Center, Winnipeg, Manitoba, Canada